CLINICAL TRIAL: NCT05372991
Title: A Two-Stage, Phase 1/2 Study to Evaluate the Safety, Tolerability and Pharmacodynamics of CBT-009 Eye Drop in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacodynamics Evaluation of CBT-009 Eye Drop
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CBT-CS201
Record Dates: First submitted 2021-05-05; First posted 2022-05-13 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-05

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.025% atropine sulphate (Active Comparator): The comparator formulation of 0.025% atropine sulfate monohydrate in normal saline will be prepared by diluting commercial 1% atropine sulphate solution with physiologic saline.
  Interventions: Drug: Atropine Sulfate
- vehicle (Placebo Comparator): CBT-009 vehicle formulation is a proprietary sterile ophthalmic solution that does not contain CBT-009 drug substance.
  Interventions: Drug: Vehicle
- CBT-009, Low Dose (Experimental): CBT-009 low dose formulation is a proprietary sterile ophthalmic solution that contain low dose of CBT-009 drug substance.
  Interventions: Drug: CBT-009
- CBT-009, Mid Dose (Experimental): CBT-009 mid dose formulation is a proprietary sterile ophthalmic solution that contain mid dose of CBT-009 drug substance.
  Interventions: Drug: CBT-009
- CBT-009, High Dose (Experimental): CBT-009 high dose formulation is a proprietary sterile ophthalmic solution that contain high dose of CBT-009 drug substance.
  Interventions: Drug: CBT-009

INTERVENTIONS:
Drug: CBT-009 — This is a Two-Stage Phase 1/2 study to evaluate the safety, tolerability and pharmacodynamics of CBT-009 eye drop in healthy volunteers.
  Other Names: Atropine
  Arms: CBT-009, High Dose; CBT-009, Low Dose; CBT-009, Mid Dose
Drug: Vehicle — This is a Two-Stage Phase 1/2 study to evaluate the safety, tolerability and pharmacodynamics of CBT-009 eye drop in healthy volunteers.
  Other Names: Without Atropine
  Arms: vehicle
Drug: Atropine Sulfate — This is a Two-Stage Phase 1/2 study to evaluate the safety, tolerability and pharmacodynamics of CBT-009 eye drop in healthy volunteers.
  Other Names: 0.025% eyedrop aqueous solution
  Arms: 0.025% atropine sulphate

SUMMARY:
This is a Two-Stage Phase 1/2 study to evaluate the safety, tolerability and pharmacodynamics of CBT-009 eye drop in healthy volunteers.

CBT-009 has the active ingredient of atropine, which at low doses, has shown to be effective in slowing down myopic deterioration. Current atropine products are prone to degradation once the container is open to the air. ADS Pharmaceutical has developed a novel atropine formulation.

DETAILED DESCRIPTION:
Type of Study:

Stage 1: Single center, open-labeled, vehicle-controlled, single ascending dose.

Stage 2: Parallel, double-masked, randomized, vehicle-controlled with dosing once-daily in one eye.

Study Population:

Male or female healthy volunteers aged 18-36 years.

Number of Subjects and Sites:

Stage 1: Enrollment is planned for approximately 32 healthy volunteers with 8 subjects per cohort for a total of 4 cohorts.

Stage 2: Enrollment is planned for approximately 50 healthy volunteers with 25 subjects per cohort for a total of 2 cohorts.

Duration of Study Participation:

Stage 1: One day. Stage 2: 28 days of treatment with no follow-up observations.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteer without any active ocular diseases

* 18-36 years of age
* Able to provide written informed consent and comply with study assessments for the full duration of the study

Exclusion Criteria:

Uncontrolled systemic disease

* Active ocular disease
* Any ocular surgical procedure within the last 3 months
* Current enrollment in an investigational drug or device study or participation in such as study within 30 days prior to entry into this study
* Any condition or situation which, in the investigator's opinion, may put the volunteer at significant risk, may confound the study results, or may interfere significantly with the volunteer's participation in the study. Allergic or sensitive to Atropine study medication or formulation excipient
* Smoking during the study
* Female patients who are pregnant, nursing, or planning a pregnancy during the study
* Current or anticipated use of topical ophthalmic medications are prohibited during the study. Volunteers must have discontinued use of ophthalmic medications for at least 2 weeks prior to Day 1 visit

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Safety on near visual acuity | 28 days
  Near visual acuity will be assessed using best-corrected distance spectacle correction with a reduced logMAR reading chart placed at 40 cm under well-lit conditions at Day 28.
Safety on accommodation | 28 days
  The accommodation will be measured using a near point rule with best-corrected distance spectacle correction at Day 28.
Safety on mesopic and photopic pupil | 28 days
  Mesopic pupil size and photopic pupil size will be measured with a pupillometer at Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Revell, MD, Principal Investigator — University of Sunshine Coast，Australia
Locations (1):
- USC, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No